CLINICAL TRIAL: NCT00350623
Title: A Phase IIa Dose-Refinement Study of the Safety and Immunogenicity of a 3-Dose Regimen of the Merck Adenovirus Serotype 5 HIV-1 Gag/Pol/Nef Vaccine in Healthy Adults
Brief Title: Investigation of V520 in a HIV Vaccine Dose Refinement Study (V520-027)(TERMINATED)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V520-027; 2006_501
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Results first posted 2010-11-04 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infections
Keywords: AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose (Experimental): MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose (V520)
- MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose (Experimental): MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose (V520)
- MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose (Experimental): MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Interventions: Biological: MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose (V520)

INTERVENTIONS:
Biological: MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose (V520) — 3-dose regimen of 1.0-mL intramuscular injections of MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Other Names: V520
  Arms: MRKAd5 HIV-1 gag/pol/nef 4 x 10^9 Ad5 vg/dose
Biological: MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose (V520) — 3-dose regimen of 1.0-mL intramuscular injections of MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Other Names: V520
  Arms: MRKAd5 HIV-1 gag/pol/nef 8 x 10^9 Ad5 vg/dose
Biological: MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose (V520) — 3-dose regimen of 1.0-mL intramuscular injections of MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose, 3 doses administered at Day 1, Week 4, and Week 26.
  Other Names: V520
  Arms: MRKAd5 HIV-1 gag/pol/nef 1.5 x 10^10 Ad5 vg/dose

SUMMARY:
This study will test the safety and immunogenicity of an investigational Human Immunodeficiency Virus (HIV) vaccine. Immunogenicity will be measured by evaluating the immune response to several different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates good general health
* Human Immunodeficiency Virus (HIV), Hepatitis B surface Antigen (HBsAg), and Hepatitis C (HCV) seronegative
* Low risk of acquiring HIV infection
* ALT lab value within normal range

Exclusion Criteria:

* Previously received an investigational HIV vaccine
* Has a known or suspected impairment of immunologic function
* Has a clinically significant chronic medical condition that is considered progressive
* Has a major psychiatric illness
* Has any history of malignancy, with the exception of basal cell or squamous cell skin cancer
* Weighs less than 105 lbs.
* Has a recent (within two years) history of chronic alcohol abuse
* Has a contraindication to intramuscular (IM) injection, such as anticoagulant therapy or thrombocytopenia
* Female is pregnant or breast feeding, or expecting to conceive or donate eggs during the study
* Male subject is planning to impregnate or provide sperm donation during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase IIa; First Patient In: 24-Oct-2006; Last Patient Last Visit 30-May-2008. 21 sites, all in the United States of America.
Pre-assignment Details: All patients had to demonstrate good health, be at low risk of acquiring HIV infection, and met a number of laboratory criteria. They could not have previously received an investigational HIV vaccine, had a contraindication to intramuscular injection, or weighed less than 105 pounds.
Period: Overall Study
Arm/Group | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose
Started | 71 | 71 | 68
Completed | 63 | 67 | 62
Not Completed | 8 | 4 | 6
Not completed — Lost to Follow-up | 8 | 3 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — patient traveling outside the country | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose | Total
Number analyzed (Participants) | 71 | 71 | 68 | 210
Age, Continuous [Mean (Full Range); unit: years] | 30.6 [18 to 50] | 31.5 [18 to 50] | 32.0 [19 to 50] | 31.4 [18 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 38 | 37 | 106
  Male | 40 | 33 | 31 | 104
Ethnicity [Number; unit: Participants]
  Hispanic or Latino | 9 | 9 | 12 | 30
  Not Hispanic or Latino | 62 | 62 | 56 | 180
Race [Number; unit: participants]
  Asian | 1 | 2 | 4 | 7
  Black or African American | 9 | 9 | 10 | 28
  Multi-Racial | 4 | 3 | 1 | 8
  Other (Unknown) | 0 | 0 | 1 | 1
  White | 57 | 57 | 52 | 166

OUTCOME MEASURES:

1. Primary Outcome: Number of Enzyme-linked Immunosorbent Spot (ELISPOT) Responders at 30 Weeks
Time Frame: 30 weeks
Population: No data analysis was performed.
Arm/Group | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-Serious and Serious AEs were collected for 14 days following each vaccination.
Description: In addition, SAEs that occurred outside the time period specified above were collected if they were either a death or an SAE that was considered possibly, probably, or definitely vaccine related.
Arm/Group | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/71 | 2/68
Other Adverse Events (participants affected / at risk) | 56/71 | 63/71 | 60/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose (N=71) | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose (N=71) | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose (N=68)
Pyrexia (General disorders) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MRKAd5 HIV-1 Gag/Pol/Nef 4 x 10^9 Ad5 vg/Dose (N=71) | MRKAd5 HIV-1 Gag/Pol/Nef 8 x 10^9 Ad5 vg/Dose (N=71) | MRKAd5 HIV-1 Gag/Pol/Nef 1.5 x 10^10 Ad5 vg/Dose (N=68)
Eye pruritus (Eye disorders) | 2 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5
Nausea (Gastrointestinal disorders) | 4 | 9 | 5
Vomiting (Gastrointestinal disorders) | 2 | 1 | 2
Chills (General disorders) | 3 | 4 | 10
Fatigue (General disorders) | 4 | 5 | 11
Hangover (General disorders) | 0 | 0 | 3
Influenza like illness (General disorders) | 0 | 4 | 2
Injection site bruising (General disorders) | 2 | 2 | 3
Injection site erythema (General disorders) | 16 | 21 | 13
Injection site movement impairment (General disorders) | 1 | 2 | 0
Injection site pain (General disorders) | 44 | 54 | 47
Injection site pruritus (General disorders) | 2 | 4 | 1
Injection site swelling (General disorders) | 12 | 20 | 15
Malaise (General disorders) | 2 | 5 | 5
Pain (General disorders) | 1 | 6 | 7
Pyrexia (General disorders) | 3 | 9 | 13
Pharyngitis (Infections and infestations) | 2 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Dizziness (Nervous system disorders) | 3 | 4 | 5
Headache (Nervous system disorders) | 14 | 31 | 21
Lethargy (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 2 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 7 | 7
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0

LIMITATIONS AND CAVEATS:
An interim analysis of a related study, V520-023 (NCT00095576), showed that the vaccine used in V520-027 (NCT00350623) was not efficacious; therefore, vaccinations in V520-027 were stopped and only a high level summary of safety data was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.